CLINICAL TRIAL: NCT00533793
Title: A Phase II Randomized, Controlled, Open-labeled (Dose-blinded) Dose Finding Study of the Safety and Efficacy of I-040202 in the Treatment of Patients With Acute Open Tibial Shaft Fractures
Brief Title: Adjunctive Therapy to Treat Tibial Shaft Fractures
Acronym: TSF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kuros Biosurgery AG (Industry)
Collaborators: Baxter BioScience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS I-040202/01
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Trauma
Keywords: bone, tibial shaft fracture
MeSH Terms: conditions — Wounds and Injuries | interventions — Open Fracture Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SoC (Active Comparator): Standard of Care
  Interventions: Procedure: open fracture reduction
- SoC plus 0.133 mg/mL (Active Comparator)
  Interventions: Procedure: open fracture reduction
- SoC plus 0.4 mg/mL (Active Comparator)
  Interventions: Procedure: open fracture reduction
- SoC plus 1.0 mg/mL (Active Comparator)
  Interventions: Procedure: open fracture reduction

INTERVENTIONS:
Procedure: open fracture reduction — internal fracture fixation: osteosynthesis plates or intra-medullary nails

SUMMARY:
A phase 2, prospective, randomized, controlled, open-label (dose-blinded), parallel group, international multi-center study. The study will consist of four treatment groups - one control group (SoC) and three I-040202 groups receiving SoC plus 0.133 mg/mL, 0.4 mg/mL or 1.0 mg/mL I-040202.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients must meet all of the following inclusion criteria:

1. patients with an acute open fracture of the tibial shaft secondary to trauma assessed by medical examination and current radiographs indicated for open fracture reduction and internal fixation using osteosynthesis plates or intra-medullary nails
2. soft tissue management (if medically warranted, eg. debridement, irrigation, application of antibiotics) performed according to local hospital practice no later than 24h after the trauma
3. male and female patients >= 18 years
4. body mass index (BMI) 16-33 (minimum body weight 50 kg, maximum 140 kg)
5. females of child-bearing potential must be willing to undergo a pregnancy test (urine) prior to treatment start (at screening)
6. females of child-bearing potential randomized in the intervention group must agree to have acceptable contraception for at least 3 months after receiving the study medication.

   Acceptable contraceptive measures are:
   * Hormonal types of birth control with a failure rate of less than 1% per year (such as implants, injections, combined oral contraceptives, patches or other methods) or copper IUDs or other IUDs with a failure rate of less than 1% per year, AND
   * An additional barrier type of birth control measure (such as condoms, diaphragms, cervical caps, etc.) Sterilized women and abstinent women of child-bearing potential will not be required to take contraceptive measures
7. willingness and ability to understand, participate and comply with the study requirements
8. patient be able to give consent personally and sign the Informed Consent Form.

Exclusion criteria:

Patients will be not eligible if they meet one of the following exclusion criteria:

1. IIIc open fracture according to the Gustilo-Anderson classification
2. tibial defects requiring bone-grafting (e.g. large segmental defects)
3. duration from trauma to surgery longer than 14 days
4. concomitant acute bone injuries and/or major skin or other significant injuries that in the opinion of the investigator would interfere with the tibial shaft fracture healing process
5. concomitant ipsilateral tibial fractures other than in the diaphyseal region
6. evidence of immune suppression
7. suspected or known hypersensitivity to the study medication or components of it
8. evidence of hypercalcemia
9. hyperparathyroidism
10. on treatment and/or planned treatment with products containing PTH (e.g. Forteo)
11. pregnant or lactating females
12. participation in another clinical trial within the last 3 months
13. active or past history of malignant tumor
14. history or evidence for any hereditary or acquired chronic metabolic bone disease other than primary osteoporosis.
15. history or evidence for any clinically relevant organ failure or any other relevant medical condition that, in the opinion of the investigator, will relevantly interfere with the assessment of study outcome or will impose hazard to the patient if study therapy will be initiated
16. known history of allergy to anaesthetics
17. evidence of moderate or severe renal failure (serum creatinine > 3.0 times ULN, NCI CTC grades 3 and 4)
18. known history of allergic thrombocytopenia (type II) induced by heparin
19. inexplicable elevations of alkaline phosphatase or alkaline phosphatase > 5.0 times ULN, NCI CTC grades 3 and 4
20. prior external beam or implant radiation therapy to the skeleton

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2007-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Clinical Criteria:weight bearing,red.pain,walking without aid;lack of need for surg. interv. fracture site;Radiogr. crit.:Cortical bridging,disintegration/disappearance fracture lines,absence of signs for complications(infection,malunion) | short term follow-up: 6 months; long term follow-up: additional 6 months (total duration of 1 year)

SECONDARY OUTCOMES:
Prop. patients healed 3,9,12 mths after T0; prop. time, extent radiogr. union for 2,3,4,5,6,9,12 mths after T0; Eval.:6 and 12 mths; prop./invasiven. sec. interv. due to persistent non-union within 6,12 mths after T0. | short term follow-up: 6 months; long term follow-up: additional 6 months (1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Jamieson, MD, Study Director — Kuros Biosurgery
Locations (49):
- Bulgaria (2):
  - MHAT ''Sveti Georgi'', Orthopaedic and Traumatology clinic (85), Plovdiv
  - MHATEM ''N.I.Pirogov'' Second clinic of Orthopaedic and Traumatology (84), Sofia
- Czechia (2):
  - Czech Republic (51), Brno
  - Czech Republic (52), Prague
- Finland (3):
  - Finland (71), Kuopio
  - Finland (72), Oulu
  - Finland (70), Turku
- France (4):
  - France (14), Dijon
  - France (16), Dunkirk
  - France (15), Limoges
  - France (11), Rouen
- Germany (7):
  - Germany (50), Göttingen
  - Germany (43), Kiel
  - Germany (40), Leipzig
  - Germany (41), Ludwigshafen
  - Germany (44), München
  - Germany (42), Ravensburg
  - Germany (45), Rostock
- Hungary (6):
  - Fovarosi Onkormanyzat Szent janos Korhaza (81), Budapest
  - Hungary (54), Debrecen
  - Vaszary Kolos Hospital Esztergom (78), Esztergom
  - Hungary (79), Kaposvár
  - Hungary (55), Nyíregyháza
  - Hungary (53), Pécs
- Italy (21), Rozzano, Italy
- Romania (8):
  - Romania (59), Bucharest
  - Romania (58), Bucharest
  - Spitalul Universitar de Urgenta Bucuresti (87), Bucharest
  - Romania (57), Cluj-Napoca
  - Spitalul Clinic Judetean Constanta (88), Constanța
  - Romania (73), Oradea
  - Romania (74), Sibiu
  - Romania (56), Timișoara
- Serbia (5):
  - Serbia (60), Belgrade
  - Serbia (76), Belgrade
  - Serbia (61), Belgrade
  - Serbia (62), Kragujevac
  - Serbia (75), Novi Sad
- Slovakia (4):
  - Slovak Republic (65), Banska Bysterica
  - Slovak Republic (64), Bratislava
  - Slovak Republic (77), Trnava
  - Slovak Republic (63), Žilina
- Slovenia (2):
  - Slovenia (67), Izola
  - Slovenia (66), Novo Mesto
- Switzerland (5):
  - Switzerland (02), Aarau
  - Switzerland (03), Davos
  - Switzerland (01), Lausanne
  - Switzerland (04), Lucerne
  - Switzerland (05), Sankt Gallen